CLINICAL TRIAL: NCT02313558
Title: Efficacy of a Commercial Dentifrice Containing Ilex Rotunda Thunb Extract for Dental Plaque and Gingivitis: A 3-month Clinical Study in Adults in China
Brief Title: Efficacy of a Commercial Dentifrice Containing Ilex Rotunda Thunb Extract for Dental Plaque and Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: West China College of Stomatology (Other)
Responsible Party: Principal Investigator, Liu Hongchun, Ph.D., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dentifrice-36
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Gingivitis; Dental Plaque
Keywords: dentifrice; gingivitis; dental plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dentifrice Containing Ilex Rotunda Thunb (Experimental): use the dentifrice containing Ilex Rotunda Thunb to brush teeth twice daily for 12 weeks
  Interventions: Drug: Dentifrice Containing Ilex Rotunda Thunb
- control dentifrice (Placebo Comparator): use the control dentifrice to brush teeth twice daily for 12 weeks
  Interventions: Drug: Control dentifrice

INTERVENTIONS:
Drug: Dentifrice Containing Ilex Rotunda Thunb — Use the dentifrice to brush teeth twice a day for 12 weeks
  Arms: Dentifrice Containing Ilex Rotunda Thunb
Drug: Control dentifrice — Use the dentifrice to brush teeth twice a day for 12 weeks
  Arms: control dentifrice

SUMMARY:
The objective of the present study was to compare the anti-plaque and anti-gingivitis effects of a commercially available dentifrice containing 0.6% Ilicis Rotundae Cortex extract to those of a control dentifrice without any active ingredient in 12 weeks of home use.

DETAILED DESCRIPTION:
This 12-week, randomized, double-blind, parallel-group study was conducted at the State Key Laboratory of Oral Diseases, Sichuan University, Chengdu, China. The clinical study protocol and informed-consent forms were reviewed and approved by the institutional review board at the West China College of Stomatology at Sichuan University.

Prospective patients aged 18 to 70 years in good oral and general health were examined during the screening visit.Patients were included according to inclusion and exclusion criteria.

The study participants refrained from all oral hygiene procedures for at least 12 hours as well as from eating, drinking and smoking for 4 hours prior to the baseline examinations. Eligible patients were randomly assigned to receive a commercially available dentifrice containing 0.6% Ilicis Rotundae Cortex extract (experimental group) or a dentifrice without any active ingredient (control group). Random assignment to groups was performed externally by another dentist, using a computer-generated randomization sequence; all other study personnel were neither involved in the randomization process nor aware of treatment assignments in any outcome evaluation.

All dentifrices were supplied in their original packaging (the experimental and control dentifrices were identical in appearance [including size, color, and shape] and taste). The dentifrices were covered to mask their identity and provided with a unique code that was not decoded until the conclusion of the study. The test product was distributed in a separate area, and all other study personnel and study participants were blinded to treatment assignment.

Patients were provided with their assigned product and the same soft-bristled toothbrush for unsupervised brushing for 12 weeks. Patients were instructed to brush their teeth twice a day (in the morning and in the evening) for 1 minute, using enough toothpaste to cover the entire brush, and to refrain from any other oral hygiene procedures throughout the duration of the study. There were no restrictions regarding diet or smoking habits during the course of the study. Patients were requested to return to the clinic after 6 weeks and 12 weeks for follow-ups, having refrained from all oral hygiene procedures for at least 12 hours before, and from eating, drinking and smoking for 4 hours before, the scheduled visit.

Patients were evaluated at baseline, after 6 weeks, and after 12 weeks of use. At each point, patients received oral examinations of their hard and soft tissues, followed by an evaluation of gingivitis and dental plaque. Patients were asked whether they had the presence of adverse events such as any discomfort while brushing and alterations in taste. All examinations were performed by the same investigator throughout the study. However, after each examination, the gingivitis and plaque scores were kept by the facilitator, and the investigator did not have access to the scores of the patients.

Dental plaque examination: Supra-gingival plaque on the facial and lingual surfaces of each tooth was scored according to the Turesky modification of the Quigley-Hein Plaque Index.

Gingivitis examination: Gingivitis was scored according to the Löe-Silness Gingival Index.

Adverse Events: Clinical evaluations by an investigator at each scheduled visit included assessments of both oral hard and soft tissue. Patients were interviewed during these examinations for any adverse events or changes in their health status. All patients underwent their final clinical examination at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had to be aged 18 and 70 (inclusive) years in good oral and general health.
2. Patients had to possess at least 20 uncrowned permanent natural teeth (excluding third molars).
3. Patients should have a whole mouth mean plaque score of at least 1.5(Turesky modification of the Quigley-Hein Plaque Index 12-13) and a whole mouth mean gingivitis score of or greater than 1.0(Löe-Silness Gingival Index14).

Exclusion Criteria:

1. Patients were excluded from the study if they had moderate to advanced periodontal disease, 5 or more decayed untreated dental sites at screening, other disease of the hard or soft oral tissues. 2. Patients were excluded from the study if they began taking medications that can influence the study outcome, antibiotics or antimicrobial drugs, within one month prior to the start of the study or if they started taking them during the course of the study.

3. Pregnant or lactating women, patients who were participating in any other clinical study or who had participated in a study within one month prior to enrollment of study, were not allowed to participate in the study.

4. Patients were excluded from the study if they presented orthodontic bands; or partial or removable dentures; or received a dental prophylaxis anytime during the past two weeks prior to the baseline examination; or a history of alcohol or drug abuse; or used the study dentifrice within the last 3 months.

5. Patients with a history of allergies to the test products, or allergies to oral care/personal care consumer products or their ingredients, or patients with existing medical conditions, which prohibits them eating and drinking for periods up to four hours, were also excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongchun Liu, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- West China College of Stomatology, Chengdu, Sichuan, China

REFERENCES:
- [Background] Mankodi S, Chaknis P, Panagakos FS, DeVizio W, Proskin HM. Comparative investigation of a dentifrice containing triclosan/copolymer/sodium fluoride and specially-designed silica and a dentifrice containing 0.243% sodium fluoride in a silica base for the control of established supra-gingival plaque and gingivitis: a 6-month clinical study. Am J Dent. 2011 Jul;24 Spec No A:21A-27A. PMID 22216654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment began in March,2013,at West China College of Stomatology Chengdu, Sichuan, China.
Pre-assignment Details: In the experimental group, 2 patients withdrew immediately after randomization; the withdrawal was not the result of the dentifrices used.
Period: Overall Study
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Started | 50 | 50
Completed | 44 | 46
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.16 (7.9) | 31.26 (7.86) | 30.72 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  China | 44 | 46 | 90
baseline dental plaque score [Mean (Standard Deviation); unit: units on a scale] — Plaque were scored at the disto-, mid-, mesio-buccal and disto-, mid-, mesio-lingual surfaces of each tooth according to the criteria of the Turesky modification of the Quigley-Hein Plaque Index: 0 =No plaque; 1 =Separate flecks of plaque at the cervical margin; 2 =A thin, continuous band of plaque (up to 1 mm) at the cervical margin; 3 =A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth; 4= Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth;5 =Plaque covering 2/3 or more of the side of the crown of the tooth.
  units on a scale | 3.08 (0.59) | 3.05 (0.46) | 3.07 (0.53)
baseline gingivitis score [Mean (Standard Deviation); unit: units on a scale] — The degree of gingivitis was scored at 6 sites (disto-, mid-, mesio-buccal and disto-, mid-, mesio-lingual) of each tooth according to the criteria of the Löe-Silness Gingival Index: 0= Absence of inflammation; 1 =Mild inflammation-slight change in color and little change in texture; 2=Moderate inflammation-moderate glazing, redness, edema and hypertrophy; 3=Severe inflammation-marked redness and hypertrophy. Tendency for spontaneous bleeding.
  Whole-mouth mean plaque scores were calculated by summing all scores for all sites and dividing by the total number of sites scored.
  units on a scale | 1.32 (0.25) | 1.35 (0.24) | 1.34 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Assessment After 6 Weeks of Dentifrice Use
Description: After 6 weeks supra-gingival plaque on the facial and lingual surfaces of each tooth was scored according to the Turesky modification of the Quigley-Hein Plaque Index. Third molars and those teeth with cervical restorations or prosthetic crowns were excluded from the scoring procedure. Plaque was disclosed and scored on each tooth surface according to the following criteria: 0 = No plaque; 1 = Separate flecks of plaque at the cervical margin of the tooth; 2 = A thin, continuous band of plaque (up to 1 mm) at the cervical margin of the tooth; 3 = A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth; 4 = Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth; 5 = Plaque covering 2/3 or more of the side of the crown of the tooth.
  Whole-mouth mean scores were obtained by averaging the values obtained over all scoreable surfaces in the mouth.
Time Frame: 6 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Number analyzed (Participants) | 44 | 46
units on a scale | 2.98 (0.56) | 3.04 (0.47)

2. Primary Outcome: Gingivitis Assessment After 6 Weeks of Dentifrice Use
Description: After 6 weeks gingivitis was scored according to the Löe-Silness Gingival Index. Each tooth was scored on facial and lingual surfaces. Third molars and those teeth with cervical restorations or prosthetic crowns were excluded from the scoring procedure. The gingiva adjacent to each tooth surface was scored as follows: 0 = Absence of inflammation; 1 = Mild inflammation: slight change in color and little change in texture; 2 = Moderate inflammation: moderate glazing, redness, edema, hypertrophy. Tendency to bleed upon probing; 3 = Severe inflammation: marked redness and hypertrophy. Tendency for spontaneous bleeding.
Time Frame: 6 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Number analyzed (Participants) | 44 | 46
units on a scale | 1.22 (0.23) | 1.30 (0.21)

3. Primary Outcome: Plaque Assessment After 12 Weeks of Dentifrice Use
Description: After 12 weeks supra-gingival plaque on the facial and lingual surfaces of each tooth was scored according to the Turesky modification of the Quigley-Hein Plaque Index. Third molars and those teeth with cervical restorations or prosthetic crowns were excluded from the scoring procedure. Plaque was disclosed and scored on each tooth surface according to the following criteria: 0 = No plaque; 1 = Separate flecks of plaque at the cervical margin of the tooth; 2 = A thin, continuous band of plaque (up to 1 mm) at the cervical margin of the tooth; 3 = A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth; 4 = Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth; 5 = Plaque covering 2/3 or more of the side of the crown of the tooth.
  Whole-mouth mean scores were obtained by averaging the values obtained over all scoreable surfaces in the mouth.
Time Frame: 12 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Number analyzed (Participants) | 44 | 46
units on a scale | 2.53 (0.5) | 2.93 (0.44)

4. Primary Outcome: Gingivitis Assessment After 12 Weeks of Dentifrice Use
Description: After 12 weeks gingivitis was scored according to the Löe-Silness Gingival Index. Each tooth was scored on facial and lingual surfaces. Third molars and those teeth with cervical restorations or prosthetic crowns were excluded from the scoring procedure. The gingiva adjacent to each tooth surface was scored as follows: 0 = Absence of inflammation; 1 = Mild inflammation: slight change in color and little change in texture; 2 = Moderate inflammation: moderate glazing, redness, edema, hypertrophy. Tendency to bleed upon probing; 3 = Severe inflammation: marked redness and hypertrophy. Tendency for spontaneous bleeding.
  Whole-mouth mean scores were obtained by averaging the values obtained over all scoreable surfaces in the mouth.
Time Frame: 12 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Number analyzed (Participants) | 44 | 46
units on a scale | 1.13 (0.22) | 1.30 (0.23)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dentifrice Containing Ilex Rotunda Thunb | Control Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

LIMITATIONS AND CAVEATS:
The major limitation is the lack of a positive control,that is used to determine whether the dentifrice was more or less effective than it. The adoption of an inactive control is possible when the true efficacy of the dentifrice is assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No